CLINICAL TRIAL: NCT02431572
Title: A Pilot Study to Evaluate PBR PET in Brain Tumor Patients Treated With Chemoradiation or Immunotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principal Investigators, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-421
Record Dates: First submitted 2015-04-15; First posted 2015-05-01 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Intracranial Tumors; Glioblastoma; Melanoma
Keywords: Intracranial Tumors; Glioblastoma; Melanoma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Melanoma | interventions — Vaccines; Radiation; Drug Therapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metastatic Melanoma to the Brain (Cohort A) (Experimental): * Assess Inflammation (PBR PET)
  * Immunotherapy
  * Assess Inflammation (PBR PET)
  Interventions: Other: PBR PET; Biological: Cancer Immunotherapy
- Primary Brain Tumor (Cohort B) (Experimental): * Assess Inflammation (PBR PET)
  * Immunotherapy
  * Assess Inflammation (PBR PET)
  Interventions: Other: PBR PET; Biological: Cancer Immunotherapy
- Primary Brain Tumor (Cohort C) (Experimental): * Chemoradiation
  * Assess inflammation (PBR PET)
  * Follow Patients
  Interventions: Other: PBR PET; Radiation: Radiation and chemotherapy

INTERVENTIONS:
Other: PBR PET
  Other Names: PBR28
Biological: Cancer Immunotherapy — Subjects who are to be treated with immunotherapy for glioblastoma or melanoma brain metastases will be eligible for 2 of the 3 arms.
  Other Names: Checkpoint inhibition; Vaccine
  Arms: Metastatic Melanoma to the Brain (Cohort A); Primary Brain Tumor (Cohort B)
Radiation: Radiation and chemotherapy — Subjects with glioblastoma will receive or will have received treatment with chemotherapy and radiation per the standard of care.
  Other Names: Chemoradiation
  Arms: Primary Brain Tumor (Cohort C)

SUMMARY:
This research study is studying the changes in primary and metastatic brain tumor inflammation using positron emission tomography (PET) imaging using a radioactive substance called [11C] PBR28a, which is also known as peripheral benzodiazepine receptors (PBR), or PBR-PET.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention. The purpose of a pilot study is to obtain the preliminary data needed to justify performing a larger clinical trial on the effectiveness of an investigational intervention.

Standard treatment for the subjects' disease includes chemoradiation and immunotherapy.

In PET scans, a radioactive substance is injected into the body. The scanning machine finds the radioactive substance, which tends to go to cancer cells and areas of inflammation. For the PET scans in this study, the investigators are using a radioactive substance called [11C]PBR28.

The investigators would like to see if this tracer can be used to detect changes in inflammation during tumor treatment. PBR-PET scans will be performed at screening before therapy and then several weeks/months after the start of therapy, depending on the type of therapy used. No diagnostic decisions or clinical treatment decisions will be made based on any results obtained from these PET scans, and there will be no change in care. The information from these studies may help the investigators design methods that could be used in larger studies to more completely understand the role of inflammation in the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have evidence of metastatic melanoma to the brain for Cohort A or histologically confirmed GBM for Cohorts Band C.
* Those with newly diagnosed GBM but suspected to have pseudoprogression after completion of chemoradiation can enroll in Cohort C.
* Participants must have measurable brain disease, defined as at least one lesion that is 10 mm in diameter.
* Age > 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 3 months.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits

    --- OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* For Cohort A, only patients with metastatic melanoma to the brain for whom their treating physician has planned to give immunotherapy as monotherapy are eligible for this study. This can be in the setting of a clinical trial or not.
* For Cohort B, only patients with GBM for whom their treating physician has planned to give immunotherapy are eligible for this study. This can be in the setting of a clinical trial or not.
* For Cohort C, patients with newly diagnosed GBM who have completed standard temozolomide + radiation and have suspected pseudoprogression within the first 3 months of completing chemoradiation can enroll.
* Patient must be able to undergo MRI and PET scans.
* Patient must be maintained on a stable corticosteroid regimen for 5 days prior each MR-PET scan.
* High or mixed affinity binders (Ala/Ala or Ala/Thr) based on genotyping result from PBR affinity test. This blood test will be performed as part of the screening process after consent has been obtained.
* The effects of PBR on the developing human fetus are unknown. For this reason and because radiopharmaceuticals agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Radiopharmaceutical agents are known to be teratogenic.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PBR.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because PBR is a radiopharmaceutical agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to exposure of the mother to PBR, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* HIV-positive participants are excluded because their immune system is compromised and may affect the interpretation of the imaging data.
* Patients who are not suitable to undergo MRI or PET or use gadolinium contrast due to:

  * Claustrophobia
  * Presence of metallic objects or implanted medical devices in body (i.e. cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants) The craniotomy patients will all have titanium but this is MRI compatible
  * Sickle cell disease
  * Renal failure
  * Reduced renal function, as determined by creatinine clearance < 30 mL/min based on a serum creatinine level obtained within 28 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Melanoma to the Brain (Cohort A); Primary Brain Tumor (Cohort B): * Assess Inflammation (PBR PET)
  * Immunotherapy
  * Assess Inflammation (PBR PET)
  PBR PET
  Cancer Immunotherapy: Subjects who are to be treated with immunotherapy for glioblastoma or melanoma brain metastases will be eligible for 2 of the 3 arms.
- Primary Brain Tumor (Cohort C): * Chemoradiation
  * Assess inflammation (PBR PET)
  * Follow Patients
  PBR PET
  Radiation and chemotherapy: Subjects with glioblastoma will receive or will have received treatment with chemotherapy and radiation per the standard of care.
Period: Overall Study
Arm/Group | Metastatic Melanoma to the Brain (Cohort A) | Primary Brain Tumor (Cohort B) | Primary Brain Tumor (Cohort C)
Started | 1 | 1 | 9
Completed | 0 | 1 | 9
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic Melanoma to the Brain (Cohort A) | Primary Brain Tumor (Cohort B) | Primary Brain Tumor (Cohort C) | Total
Number analyzed (Participants) | 1 | 1 | 9 | 11
Age, Continuous [Median (Full Range); unit: years] | 80 [80 to 80] | 65 [65 to 65] | 58 [27 to 75] | 59 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 0 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 7 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 8 | 10
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in PBR Uptake (Changes in PBR Uptake by PET)
Description: The change in PBR uptake in arms cohorts A and B from baseline to the start of cycle 4 for metastatic melanoma patients or cycle 3 for glioblastoma patients. The 18-kDa translocator protein (TSPO) is a protein that is expressed in mitochondria and is particularly prominently expressed by activated microglia, infiltrating macrophages, and reactive astrocytes. Thus, it is a marker of neuro-inflammation. PBR28 is a second generation PET tracer that binds to TPSO. PBR28 uptake was quantified using the standardized uptake value (SUV), which is the ratio of activity per unit volume of the region of interest (ROI) compared to cerebellum. Higher values indicate increased uptake in the ROI.
Time Frame: At baseline and 3 to 4 months post baseline
Population: Only a baseline measurement was taken for the 1 patient in cohort A. Change in PBR was therefore not possible to calculate for that patient. PBR PET was only assessed once in cohort C and is reported separately.
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Metastatic Melanoma to the Brain (Cohort A) | Primary Brain Tumor (Cohort B)
Number analyzed (Participants) | 0 | 1
percent change from baseline
  Before immunotherapy |  | 1.301 [1.301 to 1.301]
  During immunotherapy |  | 1.1219 [1.1219 to 1.1219]

2. Primary Outcome: Median PBR Uptake
Description: The median PBR28 uptake as measured by positron emission tomography (PET) following chemo-radiation. The 18-kDa translocator protein (TSPO) is a protein that is expressed in mitochondria and is particularly prominently expressed by activated microglia, infiltrating macrophages, and reactive astrocytes. Thus, it is a marker of neuro-inflammation. PBR28 is a second generation PET tracer that binds to TPSO. PBR28 uptake was quantified using the standardized uptake value (SUV), which is the ratio of activity per unit volume of the region of interest (ROI) compared to cerebellum. Higher values indicate increased uptake in the ROI.
Time Frame: At the time of suspected pseudo-progression (up to 4 weeks after consent)
Measure: Median (Full Range); unit: Ratio
Arm/Group | Primary Brain Tumor (Cohort C)
Number analyzed (Participants) | 9
Ratio | 0.8172 [0.5723 to 1.1566]

ADVERSE EVENTS:
Time Frame: Adverse event data not collected
Description: Adverse event data were not collected as a part of this trial
Arm/Group | Metastatic Melanoma to the Brain (Cohort A) | Primary Brain Tumor (Cohort B) | Primary Brain Tumor (Cohort C)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT02431572/Prot_SAP_000.pdf